CLINICAL TRIAL: NCT05503160
Title: Primäres Hormon-Sensitives Mammakarzinom: Bedarfsgerechte Optimierung Der Versorgung Durch Eine Patientenzentrierte, Digitale Anwendung
Brief Title: Primary Hormone-sensitive Breast Cancer: Need-driven Health Care Improvement by Patient-centred Digital Application
Acronym: PRISMA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: Federal Joint Committee (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PRISMA
Record Dates: First submitted 2022-08-08; First posted 2022-08-16 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: New Healthcare Approach
Keywords: quality of life; adherence
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): With validated questionnaires, patient reported outcome monitoring data on quality of life, distress and therapy-adherence are collected. In case of pathologic values, the attending breast center gets advised to intervene according to individual requirements.
  Interventions: Behavioral: Intervention
- Control (No Intervention): Standard of care

INTERVENTIONS:
Behavioral: Intervention — Structured (video-)call by qualified nursing staff with breast cancer patients, with the intention to overcome side effects, distress or non-adherence to endocrine therapy.
  Arms: Intervention

SUMMARY:
The investigators designed a prospective, 2-armed, cluster-randomized multicenter clinical trial on the effect of a by a digital application triggered intervention on quality of life and therapy-adherence among breast cancer patients, compared to standard of care.

DETAILED DESCRIPTION:
With validated questionnaires, patient reported outcome monitoring data on quality of life, distress and therapy-adherence are collected. In case of pathologic values, the attending breast center gets advised to intervene according to individual requirements.

For women with breast cancer, disease and therapy come along with loss of quality of life. Therapy and its side effects often result in unauthorized discontinuation of therapy by patients. Non-adherence rates to endocrine therapy (ET) range from 31% to 73%. These patients have a poorer prognosis due to recurrence, progression and cancer deaths. Positive effects to increase therapy-adherence were shown for bidirectional communication. Furthermore the use of apps with reminder functions can increase adherence to cancer therapy. The intention within this project is to improve care of patients with primary breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* primary, hormone-sensitive breast cancer
* indication for adjuvant endocrine therapy (aromatase-inhibitor, tamoxifen, GnRH-analogue allone or in combination with tamoxifen/ aromatas inhibitor; combination of endocrine therapy with CDK 4/6-inhibitor/ antibody therapy/ radiotherapy)
* start of endocrine therapy <= 3 months ago
* patients with public health ensurance
* patients who are legally competent and able to understand and follow instructions of the study staff
* present informed consent

Exclusion Criteria:

* no use of internet or digital applications
* advanced, metastatic breast cancer
* simultaneous serious disease
* life expectancy < 2 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Quality of Life (QOL) | 24 Months
  Change in EORTC QLQ-C30 subscale

SECONDARY OUTCOMES:
Quality of Life (QOL) | 24 Months
  Change in EORTC QLQ-BR23
Quality of Life (QOL) | 6, 12, 18 Months
  Change in EORTC QLQ-BR23
Quality of Life (QOL) | 6, 12, 18 Months
  Change in EORTC QLQ-C30
Adherence | 24 Months
  Number of days missing tablets
Mental health | 24 Months
  Change in GAD-2
Mental health | 24 Months
  Change in Distress thermometer
Mental health | 24 Months
  Change in PHQ-2
Adverse effect of therapy | 24 Months
  Count of side effects cat. 3/4
Assessment of new digital form of care | 24 Months
  Usefulness of application
Progression free survival | 24 Months
  PFS rate
Overal survival | 24 Months
  OS rate
Total cost | 24 Months
  Cost difference
Disease-specific costs | 24 Months
  Cost difference
Effectiveness (QOL) | 24 Months
  Change in EORTC QLQ-C30 subscale
Efficiency (QALY) | 24 Months
  Qaly-Index from EQ-5D-5L
Patient Satisfaction | 6, 24 Months
  Short Assessment of Patient Satisfaction - Satisfaction Index
Stakeholder perspective | 12, 24 Months
  Stakeholder perspective questionnaires
Number of Interventions | 24 Months
  Automatically initiated reasons for interventions

CONTACTS AND LOCATIONS:
Overall Officials: Marion Kiechle, Prof. Dr. med., Study Director — Technical University of Munich
Locations (1):
- Klinikum rechts der Isar, Frauenklinik, Technische Universität München, Munich, Germany, Germany